CLINICAL TRIAL: NCT00832741
Title: Secretion and Significance of the Incretin Hormones on the Postprandial Glycemic Response in Type-1 Diabetes Mellitus
Brief Title: Incretin Hormones in Type-1 Diabetes Mellitus Glycemic Response in Type-1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Urd Kielgast, MD, Hvidovre University Hospital
Other Study IDs: H-C-2007-0080; 2008-41-1811
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Type 1 Diabetes
Keywords: GLP-1; Type 1 diabetes; Glycemic control; Incretin hormone
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — whole blood, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate whether secretion of incretin hormones is intact and to what extent endogenous as well as exogenous GLP-1 controls postprandial glucose excursions in patients with type-1 diabetes mellitus.

DETAILED DESCRIPTION:
GLP-1 and GIP are incretin hormones secreted from specific endocrine celles in the gut. Stimulus for secretion is prescence of carbohydrates, fat and protein in the gut. The incretin hormones controls postprandial glucose excursions through stimulation of insulinsecretion as well as inhibition of glucagon and gastric emptying.The effects of GLP-1 on insulin secretion and glucagon inhibition are glucose dependent and the risc of hypoglycemia is therefore negligible when the hormone is administered in supra physiological concentrations.Furthermore, some animal studies suggest that GLP-1 has a trofic effect on the betacells and the hormone has been shown to replenish intracellular stores of insulin. Because the main bloodglucose lowering effect of GLP-1 has been thought to be due to increased insulin secretion, analouges of the hormone has been developed for the treatment of type-2 diabetes. So far, relatively little is known about the effect of GLP-1 in type-1 diabetes.It possible, that GLP-1 in combination with insulin (possibly mainly through its effect on glucagon inhibition and gastric emptying) could reduce the need for exogenous insulin with a concomitant reduced risc of hypoglycemia. Without compromising the target glucemic control. This study focuses of the postprandial bloodglucose lowering effects of endogenous as well as exogenous GLP-1 in patients with type-1 diabetes according to residual betacell function and glycemic control.Furthermore, the endogenous secretion of incretin hormones in patients with type-1 diabetes mellitus will be compared to that of matched normal controls.

ELIGIBILITY:
Inclusion Criteria:

* type-1 diabetes mellitus
* diagnosis between 5-40 years.
* age 18-60 year
* normal weight at time of diagnosis
* insulintreatment from diagnosis
* HbA1c < 7.6 %

Exclusion Criteria:

* diabetic complications
* disease other than type-1 diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic patients and community population(control subjects)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
blood glucose | 4 hours

SECONDARY OUTCOMES:
GLP-1 and GIP response during a meal | 4 hours
betacell function (incremental area under the c-peptide concentration curve) | 4 hours
alfa cell function (plasma glucagon) | 4 hours
gastric emptying | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Urd Kielgast, MD, Study Director — unafilliated; Sten Madsbad, MD, DMSc, Principal Investigator — Unafilliated
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark